CLINICAL TRIAL: NCT06147804
Title: Managment and Outcome of Urinary Bladder Trauma After Gynaecological and Obstetric Operations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ashraf Abdelmageed Hamdallah, Resident, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UB trauma after gyn&obs op
Record Dates: First submitted 2023-11-09; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Urinary Bladder Trauma
Keywords: Urinary bladder trauma after gynaecological and obstetric operations
MeSH Terms: interventions — Obstetric Surgical Procedures

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Females after gynaecological and obstetric operations (Experimental): Comaprison of the outcome
  Interventions: Procedure: Surgical managment of Urinary bladder trauma after gynaecological and obstetric operation

INTERVENTIONS:
Procedure: Surgical managment of Urinary bladder trauma after gynaecological and obstetric operation — How to manage Urinary bladder trauma after gynaecological and obstetric operations by the best method to prevent the occurrnce of vesicouterine fistula

SUMMARY:
We aimed to evaluate the management and outcome of bladder trauma after gynecological and obstetric operations at Assiut university hospital and to evaluate the methods of treatment of these complications.

We aimed to find out risk factors for vesico uterine fistula after bladder trauma

DETAILED DESCRIPTION:
The female genital and urinary systems are closely related embryologically and anatomically. The surgeon should know the anatomy of this area to avoid urinary tract (UT) injuries during obstetric (Obst) and gynecologic (Gyn) surgeries (Solyman et al., 2022)

UT injuries during Obst/Gyn surgeries are rare but have a significant psychological impact on both patient and surgeon, and their medico legal aspects are very bothering (Safrai et al., 2022)

UT injuries during Obst/Gyn operations range from 0.3 to 1% (Blackwell et al., 2018) Most cases are bladder injury, approximately three times more than ureteral injury (Wong et al., 2018)

The primary goal of the Obst/Gyn surgeon is to avoid UT injuries during his procedure. Still, in some situations, this will be difficult as in patients with abnormal anatomy, difficult operations as in the presence of severe bleeding or pelvic adhesions, and with surgeons with low experience. Immediate intraoperative repair of these injuries is optimal. In some cases, diagnosis and management are delayed postoperatively(Patel and Heisler, 2021)

UT injuries during Obst/Gyn operations are either acute injuries such as bladder and ureteral laceration, and ureteral ligation identified immediately intra operatively or chronic injuries as fistula formation and stricture ureter, which are discovered later on (Lee et al., 2012) Iatrogenic urological complications from gynecological surgery can be prevented and reduced by complying with standard surgical

ELIGIBILITY:
Inclusion Criteria:

-

All patients with Urinary bladder injuries related to Obst/Gyn operations

Exclusion Criteria:

* no exclusion criteria in all patients with bladder trauma after gyn &obs operations

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
To measure the surgical managment of the bladder tear | Follow up after 3 weeks and 3 months and 6 months
  By the occurrence of vesicogenital fistula or not
  evaluate the prevalence of vesicogenital fistula after bladder trauma after gynaecological and obstetric operations

SECONDARY OUTCOMES:
To evaluate the quality of life, satisfaction of patients, UTI manifestations | After 3 weeks and 3 months and 6 months
  By directly questioning the patient